CLINICAL TRIAL: NCT05908019
Title: The Effects of Pulmonary Hypertension Web-Based Health Care Program on Symptom Management, Social Support, Activity Tolerance, and Quality of Life in Patients With Pulmonary Hypertension.
Acronym: PAH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Defense Medical Center, Taiwan (Other)
Responsible Party: Principal Investigator, Miao-Yi Chen, Principal Investigator, National Defense Medical Center, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: NDMC
Record Dates: First submitted 2023-06-01; First posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Web-based Health Care Program

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Web-based health care program (Experimental): We aim to develop a PAH web-based health care program, and to evaluate the effects of this program on ameliorating social support, self-care ability and active tolerance, and improving symptom distress, anxiety, depression and quality of life in patients with PAH.
  Interventions: Other: Web-based health care program
- Usual care (No Intervention): usual care

INTERVENTIONS:
Other: Web-based health care program — According to the participants' feedback and recommends, we will modify this program to make it more suitable.
  In the second and third years, we will conduct a parallel-group, double blind, and block randomization, experimental design study to examine the effectiveness of the Pulmonary Hypertension Web-Based Care Program on the improvements of patients' social support, self-care ability, active tolerance, symptom distress, depression, anxiety and quality of life in patients with PAH.
  Arms: Web-based health care program

SUMMARY:
Pulmonary arterial hypertension (PAH) is a chronic disease characterized by an elevation in pulmonary artery pressures and pulmonary vascular resistance. The condition most often is rarely detected, and patients frequently suffer symptoms for several years before being appropriately diagnosed. Patients with PH suffer from several symptoms, such as exertional dyspnea, fatigue, weakness, chest pain, fainting…et al. Pulmonary hypertension is an incurable and progressive disease with complex symptoms and treatments. Patients must learn to deal with their unpredictable future and manage the complex treatments associated with severe adverse effects and need significant changes in lifestyle.

Therefore, it is important to assist patients to develop the ability of symptom management.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years old, diagnosed by clinical specialists as patients with pulmonary hypertension (Group1 and Group 4)
2. Clear consciousness, able to communicate in Mandarin and Taiwanese, with normal hearing
3. Those who have internet or mobile internet at home
4. Adults without mental illness
5. No alcohol or drug abusers.

Exclusion Criteria:

1. critical disease

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Arterial Hypertension Symptom | Change from Baseline pulmonary Arterial Hypertension Symptom at six months
  Pulmonary Arterial Hypertension Symptom Interference Scale, PAHSS, The 10-point Likert scale higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Social support | Change from Baseline social support at six months
  Multidimensional Scale of Perceived Social Support, (MSPSS). The 7-point Likert scale higher scores mean a better outcome.This instrument is 12 questions long and has been widely used and well validated.
Activity ability | Change from Baseline activity ability at six months
  6 Minute walk test, 6MWD
Pulmonary Hypertension Quality of life | Change from Baseline quality of life at six months
  The Cambridge Pulmonary Hypertension Outcome Review, (CAMPHOR). The 5-point Likert scale higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided